CLINICAL TRIAL: NCT02921503
Title: Impact of a Mobile App on Topical Corticosteroid Prescribing by Family Practitioners
Brief Title: Topical Corticosteroid App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Joslyn S. Kirby, Associate Professor, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 00005201
Record Dates: First submitted 2016-09-29; First posted 2016-10-03 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Topical Corticosteroid, Topical, Medication, Utilization
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Topical Corticosteroids App Users (Experimental): Practitioners will asked to use a novel application during their patient encounters over the next three months. This application should not modify treatment, it will only act as a vehicle to present evidence based research. Patients will not be subjects of this research, as the app is only presenting best practice which the physicians should be aware of.
  Interventions: Other: mobile topical corticosteroid app

INTERVENTIONS:
Other: mobile topical corticosteroid app — app used on mobile phones that takes the input of providers and suggests topical corticosteroids with specific information on the ingredient, vehicle, and amount

SUMMARY:
The study aims to evaluate the effectiveness of a mobile application to assist in the prescription of topical corticosteroids (TCS), focusing on best fit choices of potency, vehicle and volume. The mobile application will be developed from the results obtained in a systematic literature review and quality assessment of clinical practice guidelines for topical corticosteroid use. The quality of the guidelines will be assessed using the AGREE II tool. After the app user enters in information concerning patients' rash location and desired treatment duration, the app will generate a list of recommended topical steroids (focusing on specific quantity and potency) for the patient's particular area of need. The objective of the study is to evaluate whether the use of a standardized application will change prescribing practices for primary care physicians, physician assistants and nurse practitioners.

DETAILED DESCRIPTION:
Primary Study Endpoints The primary endpoint of this study to be measured would be topical steroid prescription records (including unit sizes, potencies, and number of prescriptions) from study participants before and during use of this app.

Secondary Study Endpoints The study participants will also be asked to take surveys to rate user satisfaction and clinical utility.

2.1 Scientific Background and Gaps The literature has shown that patients with dermatologic conditions may not receive appropriate management by PCPs. Dermatologic conditions are common, affecting 20-36% of patients in PCP offices; however PCPs report diagnostic and management uncertainty.1,2 PCPs have been shown to prescribe either inappropriately high-potency TCS or, conversely, inappropriately low-potency TCS.3 In addition, it was recently found that drug costs may be higher if multiple small tubes are dispensed over the treatment course.4 Thus, there are opportunities to reduce cost by prescribing larger units, when indicated; however PCPs may not have the knowledge to effectively and cost-efficiently prescribe TCS. Teaching this information is not sufficient, since most (71%) medical schools provided nine or fewer hours of instruction in the first two years.5 Importantly, mobile devices and apps provide significantly increased access to point-of-care tools and, with use by providers, demonstrate better clinical decision-making and improved patient outcomes.6,7 Thus, our goal is to develop a point-of-care decision support app to educate PCPs while facilitating evidence-based care and lower health care costs.

The mobile application will be developed by a team at Penn State Hershey from the results obtained in a systematic literature review and quality assessment of clinical practice guidelines for topical corticosteroid use. The quality of the guidelines will be assessed using the AGREE II tool. After the app user enters in information concerning patients' rash location and desired treatment duration, the app will generate a list of recommended topical steroids (focusing on specific quantity and potency) for the patient's particular area of need. It is ultimately up to the physician whether or not to follow or modify the recommended suggestions.

Study Rationale Smartphone applications are rising rapidly in popularity in the healthcare field. 85% of clinicians are reported as owners of smart phones, with 50% of them using apps in their practice.8 Use of smartphone technology and clinical decision support tools may mean improvements in primary care practices by assisting in the standardization of the prescribing practices for TCS while allowing dermatologists more availability for patients with higher need.

ELIGIBILITY:
Inclusion Criteria:

1. Primary Care Providers in the Hershey Medical Center network:

   1. Attending physicians
   2. Physician assistants
   3. Nurse practitioners
2. 18 years of age or older
3. English speaking

Exclusion Criteria:

Those who do not fit the inclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
topical corticosteroid prescriptions | 3 months
  The primary endpoint of this study to be measured would be topical steroid prescription records (including unit sizes, potencies, and number of prescriptions) from study participants before and during use of this app.

SECONDARY OUTCOMES:
user satisfaction | 3 months
  The study participants will also be asked to take surveys to rate user satisfaction and clinical utility.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States